CLINICAL TRIAL: NCT04764019
Title: Intestinal Dysmotility in Patients With Functional Digestive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AG)56/2018
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-03

CONDITIONS: Gastrointestinal Motility Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients with chronic digestive symptoms in whom intestinal dysmotility is suspected
  Interventions: Diagnostic Test: High resolution intestinal manometry

INTERVENTIONS:
Diagnostic Test: High resolution intestinal manometry — Evaluation of intestinal manometry by the use a high resolution intestinal manometry catheter with 34 closely spaced sensors.

SUMMARY:
Automatic and non-invasive diagnostic methods based on the analysis of internal (intraluminal) and external (abdominal) images have been recently developed to measure intestinal motility. In patients with severe motor disorders, such as intestinal pseudo-obstruction, these new non-invasive techniques have shown to be equivalent to conventional intestinal manometry, the current gold-standard. However, these new techniques also detect less obvious signs of intestinal motor dysfunction, which are not detectable by conventional manometry.

High resolution manometry has been recently been applied to other parts of the digestive tract with great success, and probably will replace the actual gold-standard for intestinal motility evaluation. The investigators expect high-resolution manometry to be more sensitive than conventional manometry to the subtle motility disturbances detected by the new non-invasive techniques.

The purpose of this project is to demonstrate that intestinal motor function can be measured more sensitively and accurately using a combination of new technologies: high resolution manometry and the non-invasive diagnostic methods based on the analysis of images. The combined use of these techniques, following a step-wise algorithm, could allow to determine the mechanism, the affected regions and severity of the dysfunction in patients with intestinal dysmotility.

ELIGIBILITY:
Inclusion Criteria:

* Patients: digestive symptoms
* Healthy subjects: asymptomatic

Exclusion Criteria:

* Patients: organic disorders
* Healthy subjects: organic disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Contractile activity | 10 minutes
  Number of contractions

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Malagelada C, Karunaratne TB, Accarino A, Cogliandro RF, Landolfi S, Gori A, Boschetti E, Malagelada JR, Stanghellini V, Azpiroz F, De Giorgio R. Comparison between small bowel manometric patterns and full-thickness biopsy histopathology in severe intestinal dysmotility. Neurogastroenterol Motil. 2018 Mar;30(3). doi: 10.1111/nmo.13219. Epub 2017 Sep 22. PMID 28941004